CLINICAL TRIAL: NCT02834546
Title: Correlation Between Sorafenib Plasma Concentrations, Toxicity and Disease Control Rate in Patients Treated by Sorafenib for Hepatocellular Carcinoma
Acronym: ACTES
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/25
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; Sorafenib; Toxicity; Plasmatic concentration
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with HCC treated with sorafenib
  Interventions: Biological: Sorafenib plasma concentration 4 weeks after treatment initiation

INTERVENTIONS:
Biological: Sorafenib plasma concentration 4 weeks after treatment initiation — Sorafenib plasma concentrations will be assessed at 4, 8 and 16 weeks by high performance liquid chromatography. The pharmacology Unit of Bordeaux university hospital (Pr Molimard) is a French Center of reference for the dosage of TKI in the plasma

SUMMARY:
The aim of this pilot study is to correlate the sorafenib plasma concentration to observed toxicity and to the disease control rate in 100 patients undergoing a palliative treatment of hepatocellular carcinoma (HCC). If some correlations are observed, we will consider planning a larger interventional study to adjust sorafenib daily dose to plasma concentration.

DETAILED DESCRIPTION:
Sorafenib is the standard of care for the palliative treatment of HCC. The recommended dose of sorafenib in patients with HCC is 400 mg twice daily. Sorafenib dose-limiting toxicities include diarrhea, arterial hypertension and hand-foot syndrome. Owing a large inter-patient variability (near 50%) of sorafenib Area Under the Curve (AUC) over 12h, an over-exposure to sorafenib could explain acute toxicity. On the other hand, a suboptimal exposure could result in an insufficient anti-tumor activity as suggested by a recent study. This inter-patient variability of sorafenib pharmacokinetic is especially relevant in HCC. Indeed, most of HCC are developed on cirrhotic liver with often an impaired liver function, a decrease of albuminemia and sometimes ascitis. All these parameters are likely to impact the sorafenib pharmacokinetic. The aim of this pilot study is to correlate the sorafenib plasma concentration to observed toxicity and to the disease control rate in 100 patients.

The dose of sorafenib will be the recommended dose: 400 mg twice daily. Sorafenib daily doses will be only adjusted by the clinician on adverse event. Values of sorafenib AUC will not be transmitted to clinician.

Patients will be followed during 12 months with 5 visits: Week 4, Week 8, Week 16, Month 6 and Month 12. Adverse event related to sorafenib will be recorded and graded according to the NCI-CTC for Adverse Event during all the study period. Sorafenib plasma concentrations will be assessed at 4, 8 and 16 weeks. An additional dosage could be performed between W1 and W4, before dose modification, if a dose modification is necessary due to adverse events before W4.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years age
* Possibility of regular monitoring
* Ability to understand and willingness to sign written informed consent.
* Hepatocellular carcinoma histologically diagnosed or in case of inability to perform a histology by non-invasive radiological criteria endorsed by EASL/AASLD (a) presence of known cirrhosis and (b) identification of a focal hepatic lesion measuring at least 1cm in diameter with contrast uptake in the arterial phase and rapid wash out in the venous /late phase on two imaging techniques
* Patient not eligible for curative treatment (transplantation, resection, destruction or percutaneous chemo-embolization) or HCC still evolving after failure of a specific treatment
* ECOG ≤ 2
* Child-Pugh A or B
* Score BCLC B or C

Exclusion Criteria:

* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
* Cirrhosis CHILD C
* Score BCLC D
* ECOG > 2
* Digestive bleeding within 30 days before inclusion
* Subject has had a liver transplant or waiting for a liver transplant
* Subject previously treated with sorafenib
* Childbearing or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with HCC from 5 care centers in France for whom the indication of a first treatment with sorafenib was decided and who will be treated according to the recommendations of drug SmpC
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Adverse events related to Sorafenib needing a dose adjustment or a symptomatic medication | Up 8 weeks after sorafenib treatment introduction

SECONDARY OUTCOMES:
Adverse events notification | Week 8, 16, month 6 and 12 after sorafenib treatment introduction
Radiological response assessed by scan or MRI | Week 8, 16, month 6 and 12 after sorafenib treatment introduction
Progression-free survival time | Up to month 12 after sorafenib treatment introduction
Overall survival | Up to month 12 after sorafenib treatment introduction

CONTACTS AND LOCATIONS:
Overall Officials: Eric FRISON, MD, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique du CHU de Bordeaux
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Montpellier, Montpellier
  - CHU de Bordeaux, Pessac
  - CHU de Toulouse, Toulouse